CLINICAL TRIAL: NCT05092295
Title: Head and Intraocular Trauma Tool for the Identification of Mild Traumatic Brain Injury
Status: Active, not recruiting | Type: Observational
Sponsor: Rebiscan, Inc. (Industry)
Collaborators: Carilion Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 002_Q201535
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- TBI Patients: TBI participants 13 to 45 years of age, recruited from patients at a clinical research facility who present with head trauma. Clinical evaluation for the patient can be positive (target condition present) or negative (target condition absent) for mTBI. Enrollment is to occur within 2 weeks of the incident injury.
  Interventions: Device: Head and Intraocular Trauma Tool; Diagnostic Test: SCAT-5
- Controls: Participants should not be part of the Intended Use Population. Subjects that present to the hospital, clinic or emergency department, either as a patient or non-patient, with no history of head trauma.
  Interventions: Device: Head and Intraocular Trauma Tool; Diagnostic Test: SCAT-5

INTERVENTIONS:
Device: Head and Intraocular Trauma Tool — HITT device to scan eyes of participants up to 3 times (~45 seconds each) at time of admittance to study. Participant is to place chin in chin-rest and fixate on illuminated light on device.
  Other Names: HITT device
Diagnostic Test: SCAT-5 — Participant is to complete Step 2 (Symptom Evaluation) and Step 3 (Cognitive Screening) of SCAT-5 test.
  Other Names: Sport Concussion Assessment Tool - 5th Edition

SUMMARY:
Rebion has developed a device, the Rebion trauma tool (referred to as the head and intraocular trauma tool, or "HITT"), that detects ocular fixation and alignment using a binocular retinal scan. Preliminary data obtained from hospitalized patients with a clinically-confirmed traumatic brain injury (TBI) and uninjured controls indicates that the device can detect changes in ocular fixation, alignment, and saccades that are related to brain injury. This study seeks to evaluate the ability of the Rebion trauma tool to assess perturbations in eye movements resulting from TBI. The study will enroll 100 TBI patients and 100 controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-45 years
2. Presents to the facility within 2 weeks of head trauma
3. Able to provide informed consent

   • If minor, then able to provide parental consent and minor assent
4. Able to participate in the examination, including the ability to follow simple instructions
5. Fluency in English or Spanish

Exclusion Criteria:

1. Glasgow Coma Scale score of equal to or less than 13 at the time of study enrollment
2. Under the influence of alcohol or drugs
3. Previous eye surgery
4. Visual acuity known to be 20/200 or less in either eye
5. Known strabismus, amblyopia (lazy eye), or double vision
6. Known eye movement disorder, including nystagmus
7. Known optic nerve disease, including papilledema or optic neuropathy
8. Known retinal disease, including macular degeneration or retinal degeneration
9. Known cataract
10. History of neurosurgery
11. History of stroke/brain hemorrhage, brain tumor, or epilepsy
12. Any head trauma requiring medical attention from a physician within the last 6 months
13. Diagnosed dementia or cognitive impairment requiring assistance for daily living
14. Other condition(s) under the care of a neurologist
15. Psychiatric hospitalization in the last 90 days
16. Subject considered unsuitable for participation in this clinical trial by PI, treating clinician, or study research staff
17. Any minor brain injury regardless of loss of consciousness

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Target participants for the study population include those within 2 weeks of blunt head trauma, with a Glasgow Coma Scale score of greater than or equal to thirteen. A minimum of one hundred Target Condition subjects will be enrolled. All studies will be completed on the day of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TBI Detection | 1 day
  Patients who have diagnosed TBI and are admitted to the hospital for treatment will have their eyes scanned to identify whether the HITT device can accurately identify patients with TBI.

SECONDARY OUTCOMES:
TBI Monitor | 14 days
  Patients who have remained in the hospital for TBI and received initial HITT device scan will receive a second set of scans at 2 weeks to identify whether the HITT device can accurately identify patients with TBI.

CONTACTS AND LOCATIONS:
Overall Officials: Damon R Kuehl, MD, Principal Investigator — Carilion Roanoke Memorial Hospital
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data and individual test reports will be made available to the HITT device manufacturer to better understand its performance at identifying TBI. Personal identifiable data will not be shared with anyone outside of the Carilion Roanoke Memorial Hospital.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared on an ongoing basis, and cumulatively at the end of the study. Study length is expected to be 2 months from the first enrolled participant.
Access Criteria: Data will only be shared with researchers involved in the study at the Carilion Roanoke Memorial Hospital, and only trained staff members at the device manufacturer.